CLINICAL TRIAL: NCT07038317
Title: Identifying and Examining the Effects of Source and Presentation on Responses to Electronic Cigarette Public Education Messages in Young Adult Vapers and Non-vapers
Brief Title: A Text Messaging Trial to Test Vaping Health Messages Optimized to Young Adults' Vaping Status
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Donghee Nicole Lee, Assistant Professor, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4R00CA281094 (NIH)
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Vaping Behaviors; Message Exposure; Young Adults
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment arm will receive e-cigarette education messages with source and sidedness optimized to one's vaping status.
  Interventions: Other: Intervention
- Control (Placebo Comparator): Participants in the control arm will receive messages about sun safety.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — Intervention involves e-cigarette education messages tailored to participants' vaping status that will be sent out in SMS via text messaging three times per week over the course of 6 months.
  Arms: Treatment
Other: Control — Participants will receive non-tobacco messages (messages about sun safety) three times per week over the course of 6 months.
  Arms: Control

SUMMARY:
The goal of this study is to examine if e-cigarette education messages delivered using a source and presentation tailored to one's vaping status influences young adults' vaping behaviors. The main questions it aims to answer are:

1. Does receiving e-cigarette education messages presented using a source (expert or peer) and sidedness (one or two-sided) optimized for the current vaper group influence vaping cessation among young adults who vape daily?
2. Does receiving e-cigarette education messages presented using a source (expert or peer) and sidedness (one or two-sided) optimized for the non-vaper group influence vaping initiation among young adults who are susceptible to vaping? Participants will be randomly assigned to either the treatment (receiving messages tailored to one's vaping status) or the control (receiving non-tobacco messages) condition and receive SMS three times per week over the course of 6 months. They will complete self-report assessment and show salivary cotinine results for nicotine testing at 4 timepoints.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years old
* Fluent in English
* Not currently using tobacco products other than e-cigarettes at the time of enrollment
* Have a mobile phone to send and receive text messages

Exclusion Criteria:

* Age below 18 or above 24
* Not being fluent in English
* Currently using tobacco products other than e-cigarettes
* Not having a mobile phone

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported vaping | Baseline, six-month
  Past-30-day vaping (yes/no) will be assessed
Biochemical confirmation of vaping | Baseline, one-month, three-month, six-month
  Salivary cotinine for nicotine testing

SECONDARY OUTCOMES:
Harm perceptions | Baseline, one-month, three-month, six-month
  Participants will be asked to indicate the extent to which they think vaping nicotine (using e-cigarettes) is… safe, containing flavors that are safe to use, containing dangerous chemical, harmful to health on a scale from 1 (strongly disagree) to 5 (strongly agree).
Message perceptions | One-month, three-month, six-month
  Participants will be asked to indicate the extent to which they think the message was worth remembering, grabbed their attention, powerful, convincing, meaningful on a scale from 1 (strongly disagree) to 5 (strongly agree).
Message liking | One-month, three-month, six-month
  Participants will be asked to indicate the extent to which they liked the message they saw on a scale from 1 (dislike very much) to 5 (like very much).
Number of days of past-30-day e-cigarette use | From enrollment to the end of study at 24 weeks.
  Participants will be asked to report the number of days in the past 30 days (between 0 to 30) they used an e-cigarette.
E-cigarette accessibility | Baseline, one-month, three-month, six-month
  Participants will be assessed how they usually purchase e-cigarettes for themselves with categorical response options of…in person, from the Internet, by phone, don't buy their own. This question will only be asked if response indicates participants are between the ages of 18 and 20 AND have used e-cigarettes more than 0 days in the past 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participants dataset will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: One year after the completion of study